CLINICAL TRIAL: NCT04409431
Title: An Open-label, Cohort Study on Effects and Long-term Prognosis of Adrenal Artery Ablation and Spironolactone in Patients With Primary Aldosteronism
Brief Title: Effects of Adrenal Artery Ablation and Spironolactone in Patients With Primary Aldosteronism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA-S
Record Dates: First submitted 2020-02-10; First posted 2020-06-01 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Primary Aldosteronism; Hypertension
Keywords: Primary Aldosteronism; Hypertension; Adrenal Artery Ablation; Spironolactone
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Intervention Model Description: Patients in the Intervention group will be treated with endovascular chemical ablation of adrenal gland by endovascular injection of dehydrated alcohol. Patients in the Control group will be treated with spironolactone
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adrenal Artery Ablation (Experimental): Patients in the Intervention group will be treated with endovascular chemical ablation of adrenal gland by endovascular injection of dehydrated alcohol.
  Interventions: Procedure: Endovascular chemical Ablation of Adrenal Gland
- Spironolactone (No Intervention): Patients in this group will be treated with aldosterone 20-80mg daily according to blood pressure

INTERVENTIONS:
Procedure: Endovascular chemical Ablation of Adrenal Gland — Patients in this group will be treated with partial ablation of adrenal gland by endovascular injection of dehydrated alcohol
  Arms: Adrenal Artery Ablation

SUMMARY:
Primary aldosteronism (PA) is one of the most common cause of endocrine and resistant hypertension. Current studies have shown that the activation of the renin-angiotensin-aldosterone system (RAAS) and the increased sympathetic nerve activity in the central or local tissue are the key mechanisms of high blood pressure and its organ damages.

Current guidelines suggest that surgery and aldosterone receptor inhibitors are the only treatment for primary aldosteronism. However, only about 35% of aldosterone tumors and a small number of unilateral adrenal hyperplasia can be treated surgically. More than 60% of primary aldosteronism and bilateral adrenal hyperplasia need long-term oral aldosterone receptor inhibitors. At present, spironolactone is the most commonly used aldosterone receptor inhibitor. Long term use of spironolactone may cause hyperkalemia, hyperplasia of male mammary gland, hairiness of female and other adverse reactions. Therefore, the researchers suggest that partial removal of adrenals can reduce aldosterone level, lower blood pressure and restore potassium metabolism balance.

In patients with primary hyperaldosteronism, the level of aldosterone increases, which can cause vascular endothelial dysfunction, myocardial injury and ventricular fibrosis. The study shows that long-term oral administration of spironolactone can reverse the above cardiovascular damage and correct heart failure. Adrenal artery ablation can reduce aldosterone level, but the long-term effect on cardiovascular system is unknown. In order to confirm the effect of adrenal artery ablation on blood pressure and cardiovascular system, the researchers conducted an open cohort study on patients with primary aldosteronism (including aldosterone, idiopathic aldosteronism and adrenal hyperplasia). To observe the effect of adrenal artery ablation and spironolactone on blood pressure, blood electrolyte, metabolic index, cardiovascular events and cardiovascular death risk in patients with primary aldosteronism, and to explore its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Primary Aldosteronis diagnosed by increased Renin ratio (ARR) and serum aldosterone levels ≥15 ng / dl, and confirmed by saline injection test or captopril inhibition test.
* Idiopathic aldosteronism, bilateral adrenal hyperplasia, and unilateral adrenal hyperplasia with no superior secretion confirmed with adrenal CT and adrenal venous blood (AVS).
* The patients was diagnosed with aldosteronoma or unilateral adrenal hyperplasia but refused to surgical excision.
* Signed informed consent and agreed to participate in this study.

Exclusion Criteria:

* Aldosterone cancer.
* Hyperkalemia.
* Renal failure or the following history of nephropathy: serum creatinine 1.5 times higher than the upper limit; dialysis history; or nephrotic syndrome.
* Secondary hypertension except the primary aldosteronism.
* Adrenergic insufficiency.
* Heart failure with NYHA grade Ⅱ-Ⅳ grade or unstable angina, severe cardiovascular and cerebrovascular stenosis, myocardial infarction, intracranial aneurysm, stroke and other acute cardiovascular events.
* Acute infections, tumors and severe arrhythmias, psychiatric disorders, drugs or alcohol addicts.
* Liver dysfunction or the following history of liver disease: AST or ALT 2 times higher than the upper limit, liver cirrhosis, history of hepatic encephalopathy, esophageal variceal history or portal shunt history.
* Coagulation dysfunction.
* Pregnant women or lactating women.
* Participated in other clinical trials or admitted with other research drugs within 3 months prior to the trial.
* Any surgical or medical condition which can significantly alter the absorption, distribution, metabolism, or excretion of any study drug.
* Allergy or any contraindications for the study drugs, contrast agents and alcohol.
* Refused to sign informed consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of office systolic and diastolic pressure compared with the baseline between two groups | 3 years(End of Trial)
  Change of office systolic and diastolic pressure compared with the baseline between the intervention and control group at the end of the study
Incidence of major adverse cardiac events (MACE)(%) between two groups | 3 years(End of Trial)
  Incidence of major adverse cardiac events (MACE)(%)（cardiac death, myocardial infarction and target vessel revascularisation） between two groups at the end of the study

SECONDARY OUTCOMES:
Change of 24-h average systolic blood pressure between two groups | 3 years(End of Trial)
  Change of 24-h average systolic blood pressure between two groups at end of the study
Change of 24-h average diastolic blood pressure between two groups | 3 years(End of Trial)
  Change of 24-h average diastolic blood pressure between two groups at end of the study
Change of parameters assessed by echocardiography (IVSd、IVSs、LVPWd, LVPWs, LVEDD, LVEF, LVM) between two groups | 3 years(End of Trial)
  Change of parameters assessed by echocardiography (IVSd、IVSs、LVPWd, LVPWs, LVEDD, LVEF, LVM) between two groups at end of the study
Change of carotid intima-media thickness assessed by carotid ultrasound between two groups | 3 years(End of Trial)
  Change of carotid intima-media thickness assessed by carotid ultrasound between two groups at end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Zhu ZM, MD, Study Director — The third militery medical university
Locations (1):
- The third hospital affiliated to the Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No